CLINICAL TRIAL: NCT06578351
Title: TRacking Atopic Dermatitis Infants and Their Microbiome (TRAM)
Acronym: TRAM
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: SBB20R&33310_A
Record Dates: First submitted 2024-08-05; First posted 2024-08-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis; Pediatric ALL
Keywords: microbiome; atopic dermatitis; pediatric
MeSH Terms: conditions — Dermatitis, Atopic; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Infants: Healthy. no atopic dermatitis
- Infants with early onset of eczema: diagnosed with early onset eczema

SUMMARY:
TRacking Atopic dermatitis Infants and their Microbiome: A study to primarily assess the user experience of parents of infants with early onset eczema and parents of healthy infants on OneBiome real-world evidence research platform.

DETAILED DESCRIPTION:
Parents of healthy infants as well as parents of infants with early onset eczema:

* user experience of reading and understanding the microbiome and eating pattern analysis reports
* user experience of using and understanding the microbiome and nutrition platforms that allow parents to monitor microbiome and eating patterns of their child overtime

ELIGIBILITY:
Inclusion Criteria:

1. Infants diagnosed with early onset eczema (<12 months of age) and healthy infants (<6 months of age, before weaning).
2. Parents of children should have access to the internet and a smartphone or tablet to access the OneBiome mobile friendly website.
3. Parents of children should be able to comprehend the content in the OneBiome mobile friendly website and complete the questionnaires in English.
4. Parents of children should stay in Singapore and remain contactable.

Exclusion Criteria:

1. Children born prematurely.
2. Children with a chronic illness.
3. Children with congenital malformations, surgeries in the neonatal period or genetic syndromes.
4. Incapability of the parents of children to access OneBiome mobile friendly website and complete the questionnaires in English.
5. Any other family member is enrolled in the study.
6. Incapability of the parents of children to comply with study protocol or investigator's uncertainty about the willingness or ability of the parents of children to comply with the protocol requirements.

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants with early onset eczema (n=30, <12 months of age) and healthy infants (n=30, <6 months of age).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-01-26 (Actual); Study Completion 2026-01-26 (Actual)

PRIMARY OUTCOMES:
user experience using a survey form to evaluate user's understanding of OneBiome report | Up to age 18 months
  user experience of reading and understanding the microbiome and eating pattern analysis reports.
user experience using a survey form to evaluate user's perspective on using OneBiome report to monitor microbiome and eating pattern | Up to age 18 months
  User experience of using and understanding the microbiome and nutrition platforms that allow parents to monitor microbiome and eating patterns of their child overtime.

SECONDARY OUTCOMES:
HCP reported applicability of OneBiome concept by parents via a survey form | Up to age 18 months
  HCP reported applicability of microbiome/eating pattern profiles of their patients for their general practice, and to assess parents' overall feedback on OneBiome concept.

OTHER OUTCOMES:
Association between microbiome composition, eczema conditions and known factors that influence the microbiome in early life | Up to age 18 months
  To investigate association between microbiome composition, eczema conditions and known factors that influence the microbiome in early life including mode of delivery, antibiotic prophylaxis, infant feeding patterns and diet.
Association between microbiome composition, dietary/eating patterns, and gut health parameters | Up to age 18 months
  To determine any association between microbiome composition, dietary/eating patterns, and gut health parameters (stool consistency, frequency, colour, constipation, gastrointestinal infection, antibiotic intake) including stool images.

CONTACTS AND LOCATIONS:
Overall Officials: Bee Wah Lee, MBBS, Principal Investigator — The Child and Allergy Clinic - Mount Elizabeth Hospital; Wen Chin Chiang, MBBS, Principal Investigator — Chiang's Children Allergy and Asthma Clinic - Mount Elizabeth Hospital
Locations (1):
- Mount Elizabeth Hospital, Singapore, Singapore